CLINICAL TRIAL: NCT00804778
Title: Comparison of USCOM Cardiac Output and Continuous Thermodilution Cardiac Output in Patients With Coronary Artery Bypass Grafting
Brief Title: Comparison of USCOM Cardiac Output and Continuous Thermodilution Cardiac Output
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: department of emergency,beijing chaoyang hospital, society of emergency medicine of C.M.A
Other Study IDs: chumingyidoc@sohu.com; lcscyyy@sohu.com
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Coronary Artery Disease
Keywords: CAD; CABG; CO; CI; thermodilution; USCOM
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CABG,general anesthesia: their CO and CI was measured with USCOM and Swan-ganz cco respectively.
- group 1: co measured with swan-ganz cco combined with vigilance

SUMMARY:
It's reported that USCOM can be used to measured patients' CO and CI conveniently, accurately and not confined to place, because of it's no aggressive, it's accuracy is doubtful.

DETAILED DESCRIPTION:
18 post-CABG coronary artery disease patients receiving treatment in the SCCU of Beijing Chaoyang Hospital from March to July 2006, male (10) and female (8), with average age of 61.71士10.07 years. Aortic regurgitation or stenosis was ruled out by preoperational color ultrasonic imaging, endocardiac shunt did not exist and there was no heart valve replacement in all the patients. For all the patients after operation, pericardial cavity or left thorax close drainage, small tidal volume (6-8ml/kg) capacity controlled ventilation of breathing machine, appropriate pressure support (10-15cmH2O) and appropriate positive end-expiratory pressure were applied. Intra-aortic balloon pumping (IABP) was not used. Institutional ethics approval was obtained for the conduct of the trial.

All the patients received CABG under general anesthesia and non-extracorporeal circulation. Swan-Ganz CCO catheter (mbo 744HF75, USA) was set through right internal jugular vein or right subcalvian vein. The catheters were connected with VIGILANCE monitor after patients went back SCCU and the position of the catheters was adjusted. The bodyweight, height, instant heart rate, central venous pressure, invasive average aortic pressure and pulmonary wedge pressure of the patients were inputted into VIGILANCE monitor. VIGILANCE monitor automatically and intermittently displayed and saved the results of CO, CI, SVR, PVR and other hemodynamic parameters. VIGILANCE determined the hemodynamic parameters every 40-55seconds based on the signal noise ratio.

The period of USCOM monitoring time after CABG was 0.5-6hrs. Lowered the bed head and had the patients in horizontal position during the monitoring. Monitoring area was AV area. Turned on USCOM, selected AV mode, inputted the sex, height, bodyweight and birth date of the patients. Applied ultra transmission gel on the probe to let the probe contact the skin closely and let the probe point to the gluteal region nearly. USCOM screen automatically displayed the lateral border of the Doppler blood flow curve scanned with flow monitor and speaker displayed the acoustic signal of blood stream. The position, depth and direction of the probe were adjusted based on the figure signals and acoustic signals acquired with USCOM probe. Adjusted the sound volume, wave gain or contrast or turned the patient head gently. It indicated that the sound wave emitted by the probe had passed through aortic valve orifice or the root of aorta and the direction of sound beam paralleled to the blood flow through the aorta valve orifice when USCOM screen displayed maximum Doppler blood velocity wave and speaker displayed sharp and strong blood acoustic signals. The results were frozen and saved . Optimal measuring site, depth the probe was depressed down and direction of the probe were marked for the next measurement. Continuous 3-5 Doppler flow curves and the CO and CI measured on them were taken each time. The flow curves of one respiratory circle were taken for atrial fibrillation patients. For round probe, plane diameter was 1.5cm and frequency was 3.3MHz. The probe was disinfected with Iodophors each time before and after the measurement. The data of patient height, bodyweight and age, and operation duration was acquired from anesthesia note. CO time intervals measured with the two methods were about 2min. There was at least 30min interval between each pair of CO. Three to four pairs of CO and CI data were taken for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All 18 post-CABG coronary artery disease patients receiving treatment in the SCCU of Beijing Chaoyang Hospital from March to July 2006, male (10) and female (8), with average age of 61.71士10.07 years.

Exclusion Criteria:

* Aortic regurgitation or stenosis was ruled out by preoperational color ultrasonic imaging, endocardiac shunt did not exist and there was no heart valve replacement in all the patients.
* Intra-aortic balloon pumping (IABP) was not used.

Ages: 42 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 post-CABG coronary artery disease patients receiving treatment in the SCCU of Beijing Chaoyang Hospital from March to July 2006, male (10) and female (8), with average age of 61.71士10.07 years.For all the patients after operation, pericardial cavity or left thorax close drainage, small tidal volume (6-8ml/kg) capacity controlled ventilation of breathing machine, appropriate pressure support (10-15cmH2O) and appropriate positive end-expiratory pressure were applied. Institutional ethics approval was obtained for the conduct of the trial.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
All 18 post-CABG coronary artery disease patients receiving treatment in the SCCU of Beijing Chaoyang Hospital from March to July 2006 | The period of monitoring time after CABG was 0.5-6hrs.

SECONDARY OUTCOMES:
All 18 post-CABG coronary artery disease patients receiving treatment in the SCCU of Beijing Chaoyang Hospital from March to July 2006 | The period of monitoring time after CABG was 0.5-6hrs.

CONTACTS AND LOCATIONS:
Overall Officials: chunsheng li, professor, Principal Investigator — society of emergency medicine of C.M.A
Locations (1):
- society of emergency medicine of C.M.A, Beijing, China

REFERENCES:
- [Background] Critchley LA, Peng ZY, Fok BS, Lee A, Phillips RA. Testing the reliability of a new ultrasonic cardiac output monitor, the USCOM, by using aortic flowprobes in anesthetized dogs. Anesth Analg. 2005 Mar;100(3):748-753. doi: 10.1213/01.ANE.0000144774.42408.05. PMID 15728064
- [Background] Chand R, Mehta Y, Trehan N. Cardiac output estimation with a new Doppler device after off-pump coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2006 Jun;20(3):315-9. doi: 10.1053/j.jvca.2005.05.024. Epub 2006 Jan 18. PMID 16750729